CLINICAL TRIAL: NCT06116253
Title: Advanced Diffusion Imaging in Renal Cancer Patients: Oncologic Control and Renal Functional Reserve
Brief Title: Advanced Diffusion Imaging in Renal Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-01230
Record Dates: First submitted 2023-10-31; First posted 2023-11-03 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Renal Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Magnetic Resonance Imaging; Radionuclide Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Renal Mass Patients (Experimental): Patients will be enrolled for 2 MRI visits. These visits will include an approximately 1 hour research MRI scan and a total of between 3 and 5 hours Tc-99m DTPA scan.
  In each MRI visit, patients will be scanned for approximately one hour including both standard-of-care clinical sequences and research-based Advanced Diffusion Imaging sequences, on a Prisma 3T MRI scanner. Following the MRI exam or on a day not more than a week after the MRI exam, patients will undergo renal function assessment via Tc-99m DTPA scan and patient's kidneys will be scanned using a gamma camera. Proteinuria will be assessed by standard of care urinalysis of specimens collected at each MRI visit for each patient. Blood test will be performed at each visit to estimate GFR (eGFR) from measurement of serum creatinine.
  Interventions: Device: Magnetic Resonance Imaging (MRI) Scan; Drug: Tc-99m Pentetate

INTERVENTIONS:
Device: Magnetic Resonance Imaging (MRI) Scan — Participants will undergo a 1-hour research MRI scan.
  Other Names: Prisma 3T scanner
Drug: Tc-99m Pentetate — Participants will receive radioisotope (99mTc-DTPA) injection (5 mCi) during 3-5 hour scanning session to estimate measured glomerular filtration rate (mGFR).

SUMMARY:
The objective of this study is to apply advanced diffusion imaging in a two-pronged assessment of renal mass patients: (1) characterization of lesion malignancy and subtype, and (2) prediction of renal function stability or decline following partial nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Renal mass patients scheduled for laparoscopic partial nephrectomy.
* eGFR above 30 ml/min/m2.
* Ages 21 to 85
* Must be willing and able to provide consent.

Exclusion Criteria:

* All metal implants and dental implants that have ferromagnetic properties and are unsafe at 3.0 T.
* Pregnant women are not eligible for participating in this study.
* Acute claustrophobia

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Times Lesion Type is Correctly Predicted using IVIM-MRI at Pre-Surgery | Baseline (1 Week Prior to Operation)
  Intravoxel incoherent imaging-MRI (IVIM-MRI) data will be used to predict lesion type.

SECONDARY OUTCOMES:
Percentage of Times Post-Surgical Renal Function is Correctly Predicted Using REFMAP-MRI at Pre-Surgery | Up to Year 1 Post-Operation
  Results from the Renal Flow and Microstructure AnisotroPy-MRI (REFMAP-MRI) pre-surgical scan will be considered as predictors for either stability in renal function or incremental decline in renal function following surgery that would lead to chronic kidney disease (CKD), as defined by mGFR values and proteinuria status at follow-up.
  Post-surgical renal insult will be assessed based on either mGFR decline by over 2 ml/min/1.73 m2 per year or the appearance of proteinuria.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sigmund, PhD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This project does not contain provisions for generating public databases of anonymized individual data for future outside research. Consistent with the research plan of our funded study and the associated IRB protocol, the results of the study are made available at the aggregate level in the form of peer-reviewed publications.